CLINICAL TRIAL: NCT03225911
Title: Effect of a Lateral Wedge Insole and Simple Knee Sleeve as a Single and Combined Treatment on Biomechanical and Clinical Outcomes in Individuals With Knee Osteoarthritis (The IN-SLEEVE Study).
Brief Title: Effect of a Lateral Wedge Insole and Simple Knee Sleeve in Individuals With Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Salford (Other)
Collaborators: Northern Care Alliance NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Omar waslallah althomali, Omar Althomali, PhD student, Principal Investigator, University of Salford, University of Salford
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12345678
Record Dates: First submitted 2017-07-19; First posted 2017-07-21 (Actual); Last update posted 2017-07-24 (Actual); Status verified 2017-07

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Insole group (Experimental): This group will be treated via using lateral wedge insole. lateral wedge insole is an insole with higher lateral side than medial side. This insole is inserted in the participant shoes.
  Interventions: Device: Lateral wedge insole (insole)
- Sleeve group (Experimental): This group will be treated via using simple knee sleeve. Simple knee sleeve is a knee support which has no metal support. This sleeve is wrapped around each participant knee.
  Interventions: Device: simple knee sleeve (sleeve)
- insole + sleeve group (Experimental): this group will have treated via using the later wedge insole and the sleeve together as combined treatment. lateral wedge insole is an insole with higher lateral side than medial side. This insole is inserted in the participant shoes. Simple knee sleeve is a knee support which has no metal support. This sleeve is wrapped around each participant knee.
  Interventions: Device: simple knee sleeve + lateral wedge insole

INTERVENTIONS:
Device: Lateral wedge insole (insole) — The lateral wedge insole is an orthotic device that is placed inside the shoe. It has different thicknesses, with the lateral side being thicker than the medial side. This difference in thickness leads to the lateral side being higher than the medial side, with a different angulation.
  Arms: Insole group
Device: simple knee sleeve (sleeve) — The simple knee sleeve is support which is worn around the knee with no hinge or provide external valgus moment.
  Other Names: knee support
  Arms: Sleeve group
Device: simple knee sleeve + lateral wedge insole — The lateral wedge insole is an orthotic device that is placed inside the shoe. It has different thicknesses, with the lateral side being thicker than the medial side. This difference in thickness leads to the lateral side being higher than the medial side, with a different angulation. The simple knee sleeve is support which is worn around the knee with no hinge or provide external valgus moment.
  Arms: insole + sleeve group

SUMMARY:
The focus of this project is to determine the immediate efficacy of a combined treatment (lateral wedge insole + simple knee sleeve) in individuals with knee osteoarthritis (OA) and the short term effect over 6 weeks. Secondly, to compare the effect of this combined treatment with each treatment on its own (lateral wedge insole, simple knee sleeve)

ELIGIBILITY:
Inclusion Criteria:

* 1- Mild knee pain during walking on flat surface diagnosis via KOOS questionnaire (3 out of 10) because our aim of the study to reduce pain with combined treatment and pain lower than 3 out of 10 score might not allow to compared the pain reduction between the group.

  2- Definitive medial joint narrowing higher or equal to the lateral side and osteophytes on X-Ray A-P or PA view in weight bearing position if possible.

  3- Medial joint tenderness either by patient's indication or the clinician under the clinical examination indicating tenderness in the tibiofemoral joint.

  4- K-L grade 2 or 3 of plain radiographs. If the patient has had arthroscopy or MRI as their usual clinical care. Indication of grade 1 osteoarthritis pulse the radiological plain x-ray will be used.

  5- Being able to walk without assisted devices for 100 meters non-stop because he or she will not be able to complete this study protocol.

Exclusion Criteria:

* 1- More pain localized to patellpfemoral or lateral joint than the medial knee side on examination.

  2- Tricompartmental knee osteoarthritis. 3- K-L grade 4 or higher. 4- Neurological or orthopaedic situations known to affect the ability to walk. 5- Tibial osteotomy or any other realignment operation. 6- Total knee replacement. 7- Any condition contraindicates orthosiss (sleeve or insole) use. 8- Steroid injection to affected intra-articular knee joint space in the previous month.

  9- Previous or current use of any oththosis. 10- Participants with 30 BMI and higher will be excluded because previous study showed that individuals with 33 BMI.

  11- Lower than 35 years and higher than 85 as this period was identified to highest incidence period (Losina et al., 2013). Although individuals with 86 and higher has high prevalence to the knee OA, exclusion this population was important due to high amount of walking and balance test.

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-09-25 (Estimated); Primary Completion 2018-12-25 (Estimated); Study Completion 2019-03-25 (Estimated)

PRIMARY OUTCOMES:
External knee adduction moment (EKAM) | 6 weeks
  External knee adduction moment is a curve which is consider as indirect measurement of the knee loading. Using the gait analysis system will give us this outcome
Pain measurment. | 6 weeks
  10 cm visual analogue scale will be used to measure pain.
Muscle co-contraction | 6 weeks
  Muscle co-contraction can be measured after using Electromyography machine. This outcome gives us indicator to the effect of the treatment on muscle activity and loading.
Dynamic balance | 6 weeks
  The modified star excursion balance test will be used. In this test, the participants balance on maintaining single-leg stance, while reaching with the free limb in anterior and lateral directions in relation to the stance foot as far as they can, then return to double support without losing balance.

SECONDARY OUTCOMES:
Joint position sense | 6 weeks
  Each participant was asked to sit at the edge of a bed. Participants were blindfolded and barefoot to eliminate any other effects on the test results. After receiving instructions for the procedure and performing two practice trials, each participant was asked to extend his/her knee to one of the five randomly selected angles. The participate then will be asked to replicated the angle and the angle will be measure by using the gait lab.
Pressure pain threshold | 6 weeks
  Pressure guage will be used to measure the pain threshold on medial condyle and medial malleolus. Each participant will be asked to lie in side lying on the bed and Algometer's probe will be held perpendicular to the area which will be tested. Pain pressure threshold is defined as the lowest pressure intensity at which the pain felt. Pressure will be applied to the area tested at constant speed 10 kPa/s. each participant will be instructed to say stop when the first sensation of pain due to pressure felt. Each patient will be given 2 trials before starting the tests. Area which will be tested are the medial side of the knee as this considered the most painful area and medial malleolus as reference pain-free area (Wylde, Palmer, Learmonth, & Dieppe, 2011). Each test will be performed 3 times and the average will be calculated for each site. Pain pressure assessment will be performed at the baseline and after 6 weeks in order to investigate the treatments effect.
Physical function tests | 6 weeks
  3 functional tests will be used to investigate the effect of the treatment 40 meter fast paced walk test, 30 second chair stand test, a stair climb test).
  A- 40 meter fast paced test. Each participant will be asked to walk 10 meters' distance for 4 time which will be marked by tap on the floor.
  B- 30 second chair stand test:
  This test represents the number of counts that each participant can do to stand and sit on a chair in 30 second.
  C- 9 step stair climb test:
  In this test the time which will be taken by each participant to ascend 9 steps (20cm high) and descend will be measured in second.
Physical activity level | 6 weeks
  Exam the effect of the treatment on the physical activity level using physical activity scale for elderly questionnaire. Physical activity will be measured in this study via using physical activity scale for elderly (PASE). PASE (Appendix 7) is a valid and reliable questionnaire to measure the physical activity level (Martin et al., 1999; Ngai, Cheung, Lam, Chiu, & Fung, 2012; Washburn & Ficker, 1999).

CONTACTS AND LOCATIONS:
Overall Officials: Richard K jones, Phd, Study Director — Salford University

IPD SHARING:
Plan to Share IPD: Undecided